CLINICAL TRIAL: NCT00202683
Title: Relationship Between Succinate Dehydrogenase Mutations and High-Altitude Illness Associated With Chemoreflex Failure
Brief Title: Relationship Between Succinate Dehydrogenase Mutations and High-Altitude Illness
Status: Completed | Type: Observational
Sponsor: Société Française de Cardiologie (Other)
Other Study IDs: 2004-04
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Altitude Intolerance; High-Altitude Illness
Keywords: Altitude; Anoxemia; Mitochondria; Reflex; Genetic research
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is is the first step of a full study named CHEMOGENE because it explores the genetic determinant of an alteration of the chemoreflex. This reflex determines hyperventilation when the pressure of oxygen falls in the blood. This happens when subjects travel to high-altitude where oxygen levels diminish in the atmosphere. Subjects with such an altered chemoreflex are intolerant to altitude and develop pulmonary or cerebral edema associated with a severe headache. In this study we compare subjects tolerant to high altitude (8000 meters)to subjects intolerant to altitude. The chemoreflex is measured i.e. the hyperventilation associated with hypoxia and all subjects are scanned for the genes implicated in the mitochondrial respiratory chain. The idea is that subjects with an impaired oxygen sensing will exhibit an altered chemoreflex and will be intolerant to high-altitude.

DETAILED DESCRIPTION:
Subjects are selected at an outpatient clinic specialised in the diagnosis of tolerance to altitude, where the chemoreflex is analyzed during a bicycle exercise performed with a oxygen deprived air simulating a 8000 meters altitude.

All subjects will go later to high altitude for trekking usually. The patients are those subjects with an altered chemoreflex who exhibited cerebral edema or pulmonary edema during the trekking.

The controls are the subjects with a normal chemoreflex who did not exhibit any trouble during their journey.

Fourty subjects of each group are included. A blood sample is withdrawn and studied for succinate dehydrogenase genes in a blind fashion.

After completing the inclusion the allelic mutations will be compared in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Chemoreflex sensitivity measured (normal or pathologic)
* Journey to high-altitude (well tolerated or with a severe disease such as pulmonary edema or cerebral edema)

Exclusion Criteria:

* Asthma,
* Arterial hypertension,
* Drug treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-03; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc ELGHOZI, Prof., Principal Investigator — Institut National de la Sante et de la Recherche Medicale U 652
Locations (1):
- Centre d'Investigation Clinique, Hopital Pompidou, Paris, France

REFERENCES:
- [Background] Gimenez-Roqueplo AP, Favier J, Rustin P, Rieubland C, Crespin M, Nau V, Khau Van Kien P, Corvol P, Plouin PF, Jeunemaitre X; COMETE Network. Mutations in the SDHB gene are associated with extra-adrenal and/or malignant phaeochromocytomas. Cancer Res. 2003 Sep 1;63(17):5615-21. PMID 14500403
- [Background] Gimenez-Roqueplo AP, Favier J, Rustin P, Rieubland C, Kerlan V, Plouin PF, Rotig A, Jeunemaitre X. Functional consequences of a SDHB gene mutation in an apparently sporadic pheochromocytoma. J Clin Endocrinol Metab. 2002 Oct;87(10):4771-4. doi: 10.1210/jc.2002-020525. PMID 12364472
- [Background] Gimenez-Roqueplo AP, Favier J, Rustin P, Mourad JJ, Plouin PF, Corvol P, Rotig A, Jeunemaitre X. The R22X mutation of the SDHD gene in hereditary paraganglioma abolishes the enzymatic activity of complex II in the mitochondrial respiratory chain and activates the hypoxia pathway. Am J Hum Genet. 2001 Dec;69(6):1186-97. doi: 10.1086/324413. Epub 2001 Oct 16. PMID 11605159